CLINICAL TRIAL: NCT00863096
Title: Human Papillomavirus Screening and Vaccine Readiness Program
Status: Withdrawn | Type: Observational
Why Stopped: Unable to get the vaccine on time to offer it to the study population.
Sponsor: Public Health Research Institute, India (Other)
Collaborators: PATH (Other)
Responsible Party: Purnima Madhivanan, Public Health Research Institute
Other Study IDs: GAT.1246-04-07527-GRT
Record Dates: First submitted 2009-03-16; First posted 2009-03-17 (Estimated); Last update posted 2011-03-03 (Estimated); Status verified 2009-03

CONDITIONS: Human Papilloma Virus-Related Carcinoma
Keywords: HPV; acceptability
MeSH Terms: interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18; Papillomavirus Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Gardasil
  Interventions: Biological: Gardasil

INTERVENTIONS:
Biological: Gardasil — HPV vaccine
  Other Names: HPV vaccine

SUMMARY:
Public Health Research Institute (PHRI) is carrying out a 15 month research and advocacy project with the goals of generating critical data on acceptability, identifying determinants and facilitators of HPV vaccine uptake in adolescent girls; and investigating physicians' attitudes to identify predictors of intention to recommend immunization in Mysore, India.

DETAILED DESCRIPTION:
Discovery of the viral etiology of cervical cancer has opened up the possibility of primary prevention through vaccination. High-risk sexually transmitted types of human papillomavirus (HPV) have been identified as a necessary agent in cervical carcinogenesis, and work on vaccine development has progressed rapidly. Vaccines for HPV types 16 and 18, which are implicated in ~70% of cervical cancers, as well as types 6 and 11, which cause genital warts, have been shown to be effective and have been licensed in the last year. Modeling studies have indicated that an HPV vaccine could be cost-effective even alongside existing screening programs. Ideally, girls should be vaccinated before the onset of sexual activity, and estimates suggest that introduction of an HPV vaccination at age 12 could reduce lifetime cervical cancer incidence by up to 94%. As with any new technology, the success of HPV vaccination will be dependent on levels of acceptability and uptake. Given the need for parental consent in India, research into parental acceptance is of vital importance.

Although parental acceptance of vaccination against sexually transmitted infections (STI) including HPV, appears high in other parts of the world, there is little data in India. In previous research from other parts of the world, the biggest concern identified was that vaccinations may disinhibit risky sexual activity among adolescents. Other attitudes and beliefs that may influence parental uptake of an HPV vaccine include fear of potential side effects, concern about giving children too many vaccinations, the belief that vaccinations may cause disease, and religious and cultural taboos against vaccination. There is a critical need to develop data and experience that will provide the information needed by policymakers prior to the introduction of a cervical cancer vaccine in India.

The present research will be guided by the ecological framework and identify where the locus of HPV vaccine decision-making lies in an Indian setting. This project will explore household, peer and authority figure influencers in vaccine uptake. This process will include qualitative research methods such as focus group discussions and one-on-one interviews..

ELIGIBILITY:
Inclusion Criteria

* Potential participants must have at least one daughter between 8 and 14 years of age
* Be a decision maker for the welfare of a girl aged 8-14 years
* Be able to understand and give informed consent
* Be able to speak Kannada

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young women who participated in the formative study on acceptability of HPV vaccine in Mysore, India
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Acceptability of HPV vaccine | One year

CONTACTS AND LOCATIONS:
Overall Officials: Purnima Madhivanan Madhivanan, MD, PhD, Principal Investigator — Public Health Research Institute, India
Locations (1):
- Public Health Research Institute, India, Mysore, Karnataka, India